CLINICAL TRIAL: NCT06394219
Title: Transperitoneal Laparoscopic Pyelolithotomy: Is the Posterior Pyelotomy Better Than the Anterior? (A Randomized Controlled Clinical Trial)
Brief Title: A Comparative Study Between Anterior and Posterior Pyelotomy in Transperitoneal Laparoscopic Pyelolithotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Posterior Pyelotomy
Record Dates: First submitted 2024-04-23; First posted 2024-05-01 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Large Renal Stone
Keywords: Pyelotomy; Laparoscopic Pyelolithotomy,; pelvic stone; kidney stone
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anterior Pyelotomy (Experimental): Traditional transperitoneal laparoscopic pyelolithotomy:
  Patients who were randomized to receive classic transperitoneal laparoscopic pyelolithotomy
  Interventions: Procedure: traditional transperitoneal laparoscopic pyelolithotomy
- Posterior Pyelotomy (Experimental): Modified transperitoneal laparoscopic pyelolithotomy:
  Patients who were randomized to receive modified transperitoneal laparoscopic pyelolithotomy by applying posterior pyelotomy.
  Interventions: Procedure: modified transperitoneal laparoscopic pyelolithotomy

INTERVENTIONS:
Procedure: traditional transperitoneal laparoscopic pyelolithotomy — Performing anterior Pyelotomy.
  Other Names: TLP
  Arms: Anterior Pyelotomy
Procedure: modified transperitoneal laparoscopic pyelolithotomy — Performing posterior pyelotomy
  Arms: Posterior Pyelotomy

SUMMARY:
Large renal pelvic stones are frequently managed with percutaneous nephrolithotomy (PCNL) but laparoscopic pyelolithotomy (LPL) can be an alternative procedure when performed by skilled surgeons to achieve excellent outcomes in terms of stone free status, operative time, postoperative kidney function, hospitalization duration, and complications.

there are two methods for LPL surgery : Transperitoneal (TLP) and Retroperitoneal (RLP).

RLP associated with shorter mean time for oral intake, and mean hospital stay after surgery.

The surgical exposure in the transperitoneal route for LP is familiar to the majority of surgeons. Also, a much larger working space is available and there are various established anatomical landmarks for performing the surgery effectively. This study introduces a modified technique that creates application of posterior pyelotomy in TLP to achieve the advantages of RLP

DETAILED DESCRIPTION:
This is a randomized controlled clinical trial that aims to collect a sample within two years from the date of approval of the Scientific Research Council at Damascus University.

The study will focus on a group of patients who will undergo a transperitoneal laparoscopic pyelolithotomy surgery.

The patients will be randomly divided into two groups. The first group will undergo a traditional transperitoneal laparoscopic pyelolithotomy, which involves application of anterior pyelotomy.

The second group will receive a modified transperitoneal laparoscopic pyelolithotomy, which involves application of posterior pyelotomy.

The data will be compared between the two groups in terms of the mean duration of surgery ,mean time for oral intake ,and mean hospital stay

ELIGIBILITY:
Inclusion Criteria:

* Patients with large renal pelvic stone > 2 cm .
* failure of minimally invasive approaches such as PCNL or ESWL
* stones that were neither amenable to ESWL nor were ideally suitable for PCNL
* Patient's preference for a quick one-stage procedure.
* Negative urine culture

Exclusion Criteria:

* Patients refusing study participation.
* Contraindication to general anesthesia.
* Contraindication to laparoscopic surgery.
* Patients with an intrarenal pelvis.
* Previous surgical on the same kidney.
* Associated anatomical deformity.

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Operative time | at the end of surgery in the operating room
  the duration of the surgical procedure. It is measured by minutes, and calculated from establishing the pneumoperitoneum until the surgery is completed by suturing the skin.
  It will be measured in the outcome by the mean
Days for oral intake | Up to one week after surgery
  the number of days to start introducing oral fluids and food after surgery with good acceptance, and without vomiting or flatulence.
  It will be measured in the outcome by the mean
Days of hospital stay | up to ten days after surgery
  the number of days the patient stayed in the hospital after surgery. It will be measured in the outcome by the mean
Postoperative urine leak | up to three days after surgery
  considered to be present when the drain contained >30 cc of urine the morning after surgery.
  It is measured by answering the question: Is there any urinary leakage, yes or no? It will be measured in the outcome by the ratio
stone-free status | Up to one week after surgery
  postoperative radiological imaging demonstrating evidence of residual stones It will be measured in the Outcome by the ratio

CONTACTS AND LOCATIONS:
Locations (1):
- Damascus University, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Soltani MH, Hossein Kashi A, Farshid S, Mantegy SJ, Valizadeh R. Transperitoneal Laparoscopic Pyelolithotomy versus Percutaneous Nephrolithotomy for Treating the Patients with Staghorn Kidney Stones: A Randomized Clinical Trial. Urol J. 2021 Dec 20;19(1):28-33. doi: 10.22037/uj.v18i.6831. PMID 34927230
- [Background] Bai Y, Tang Y, Deng L, Wang X, Yang Y, Wang J, Han P. Management of large renal stones: laparoscopic pyelolithotomy versus percutaneous nephrolithotomy. BMC Urol. 2017 Aug 31;17(1):75. doi: 10.1186/s12894-017-0266-7. PMID 28859655
- [Background] Al-Hunayan A, Abdulhalim H, El-Bakry E, Hassabo M, Kehinde EO. Laparoscopic pyelolithotomy: is the retroperitoneal route a better approach? Int J Urol. 2009 Feb;16(2):181-6. doi: 10.1111/j.1442-2042.2008.02210.x. Epub 2008 Dec 2. PMID 19183229
- [Background] Gaur DD, Agarwal DK, Purohit KC, Darshane AS. Retroperitoneal laparoscopic pyelolithotomy. J Urol. 1994 Apr;151(4):927-9. doi: 10.1016/s0022-5347(17)35124-8. PMID 8126827
- [Background] Radfar MH, Dadpour M, Simforoosh N, Basiri A, Nouralizadeh A, Shakiba B, Valipour R, Zare A. Laparoscopic pyelolithotomy in patients with previous ipsilateral renal stone surgery. Urologia. 2021 Feb;88(1):41-45. doi: 10.1177/0391560319890993. Epub 2019 Dec 23. PMID 31868562
- [Background] Wang X, Li S, Liu T, Guo Y, Yang Z. Laparoscopic pyelolithotomy compared to percutaneous nephrolithotomy as surgical management for large renal pelvic calculi: a meta-analysis. J Urol. 2013 Sep;190(3):888-93. doi: 10.1016/j.juro.2013.02.092. Epub 2013 Feb 27. PMID 23454154